CLINICAL TRIAL: NCT05001607
Title: A Novel Method of Lung Isolation Compared With Standard Methods in a Model of Massive Pulmonary Hemorrhage.
Acronym: BloodyBlocker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, F. Robert Purdy, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H20-00662
Record Dates: First submitted 2021-07-30; First posted 2021-08-12 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hemorrhage
Keywords: simulation; anesthesia

STUDY DESIGN:
Intervention Model Description: Recruited anesthesiologists will sequentially perform all four methods of pulmonary blockade on an intubating manikin. The method order will be randomized to control for a learning effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study trial (Other): All participants will perform pulmonary blockade on an intubating manikin using 4 different methods: Endobronchial intubation with an endotracheal tube; Bronchial blocker attached to the outside of an endotracheal tube; Double lumen endotracheal tube; and Intraluminal placement of bronchial blocker.
  Interventions: Device: Bronchial Blocker

INTERVENTIONS:
Device: Bronchial Blocker — Trial of four methods of pulmonary blockade; one novel method and three published methods.
  Other Names: Arndt Endobronchial Blocker; Double lumen tube; Endotracheal tube

SUMMARY:
Dr. Purdy has developed a novel bronchial blocker device that has multiple applications. In this project, a simulation model of massive pulmonary hemorrhage in an adolescent intubating manikin will be used to compare the novel method against 3 published methods of lung isolation.

DETAILED DESCRIPTION:
Purpose: To compare a novel airway device in a realistic adolescent airway model of massive pulmonary hemorrhage to three standard methods of lung isolation.

Hypothesis: The novel method will be as fast or faster than traditional methods.

Justification: Lung isolation in massive pulmonary hemorrhage is associated with mortality rates as high as 40%. Current methods of lung isolation are challenging and have a number of limitations. The development of this novel device was a response to the limitations of current solutions and could significantly increase the speed and ease of placing a bronchial blocker under these circumstances.

Objectives: (1) To determine the length of time required for successful lung isolation in each of the four methods trialed. (2) To determine the length of time required for intubation in each of the four methods trialed. (3) To describe challenges in each method within the scenario of massive pulmonary hemorrhage. (4) To assess the utility of the model of massive pulmonary hemorrhage in future simulations.

Research Design: We propose a within-subject randomized procedure evaluation study comparing the placement of a novel bronchial blocker with three standard methods of lung isolation in a massive pulmonary hemorrhage simulation.

Analysis: Mixed effects model will be used to test the difference in total time to lung isolation between the novel method and the other three methods, with the subject as the random variable. If normality and homogeneity assumptions of the mixed-effects model are not fulfilled, then the non-parametric Wilcoxon signed-rank test would be used to compare the novel method to each of the other methods. Time constraints are placed on completion of a task, as such, we will complete sensitivity analysis where we include all participants in the analysis compared to excluding those that were unable to complete at least 1 method.

ELIGIBILITY:
Inclusion Criteria:

* Practicing anesthesiologists
* Anesthesia fellows

Exclusion Criteria:

* Those who don't want to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Total time to successful lung isolation. | Within 10 minutes from start of direct laryngoscopy
  Total time from start of direct laryngoscopy to establishment of lung isolation confirmed by one lung ventilation.

SECONDARY OUTCOMES:
Time to successful intubation | Within 10 minutes from start of direct laryngoscopy
  Time from the start of direct laryngoscopy to successful intubation confirmed by ventilation of both lungs.
Time to successful method placement | Within 10 minutes from successful intubation
  Time from successful intubation to establishment of lung isolation.
Model utility | At the end of the trial, within an hour of starting the first practice intubation.
  Responses on post-study questionnaire for future utility of the model in simulations, based on the Lung Isolation Techniques Simulation Training Evaluation Questionnaire (LITSTEQ) developed by Failor and colleagues (2014) https://doi.org/10.1053/j.jvca.2013.07.015, modified to specify training for massive pulmonary hemorrhage.
  Graded on a Likert scale of 1-5; 1 - Strongly disagree, 2 - Disagree, 3 - Neutral, 4 - Agree, 5 - Strongly Agree. Higher scores relate to a more positive outcome in assessing the utility of using the simulation model for massive pulmonary hemorrhage training.

CONTACTS AND LOCATIONS:
Overall Officials: F Robert Purdy, FRCA, Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No